CLINICAL TRIAL: NCT02174653
Title: Safety and Intake Effect of EPs® 7630 (an Extract of the Roots of Pelargonium Sidoides) A Prospective, Monocentric, Randomised, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Safety and Intake Effect of EPs® 7630 (an Extract of the Roots of Pelargonium Sidoides)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Willmar Schwabe GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 701079.01.013; 2013-004977-28 (EudraCT Number)
Record Dates: First submitted 2014-06-02; First posted 2014-06-25 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold | interventions — Desiccation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- EPs® 7630 (Active Comparator): Active Comparator 20 mg EPs® 7630 film-coated tablet
  * During the common cold free period: One film-coated tablet (20 mg) three times a day
  * During a common cold episode: Two film-coated tablets (1 x 20 mg and 1x placebo) three times a day (in the morning, midday and evening; total daily dose 60 mg) over the individual treatment duration of 14 consecutive days.
  Interventions: Drug: EPs® 7630; Drug: Placebo
- EPs(R) 7630 (Active Comparator): Active Comparator 20 mg EPs® 7630 film-coated tablet
  * During the common cold free period: One film-coated tablet (20 mg) three times a day
  * During a common cold episode: Two film-coated tablets (2 x 20 mg = 40 mg) three times a day (in the morning, midday and evening; total daily dose 120 mg) over the individual treatment duration of 14 consecutive days.
  Interventions: Drug: EPs® 7630
- Placebo (Placebo Comparator): * During the common cold free period: One film-coated tablet (placebo) three times a day
  * During a common cold episode: Two film-coated tablet (placebo) three times a day (in the morning, midday and evening) over the individual treatment duration of 14 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EPs® 7630 — 20 mg EPs® 7630 film-coated tablets during 4 months Orally intake three times a day (in the morning, midday and evening)
  Other Names: Pelargonium root liquid extract, dried
  Arms: EPs(R) 7630; EPs® 7630
Drug: Placebo — Control: Placebo film coated tablets during 4 months Orally intake three times a day (in the morning, midday and evening)
  Arms: EPs® 7630; Placebo

SUMMARY:
The aim of the study is to evaluate the safety of the intake of EPs® 7630 during a long-term (4 months) medication. The protective effects of EPs®7630 and its effects during a cold episode will also be studied.

DETAILED DESCRIPTION:
The main objective of this clinical trial is to evaluate the safety of EPs® 7630 intake - used as continuous protection and at the onset of cold symptoms - in adult participants during a long-term (4 months) medication. Due to the sparseness of empirical data in the population and this setting, no confirmatory hypotheses are formulated and the data will be analysed descriptively.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female participant (at least 18 years old)
2. Participant provided a written informed consent in accordance with the legal requirements
3. Participant with willingness and ability to comply with all procedures of the clinical trial and be available for the duration of the study
4. Participant is of good physical and mental condition
5. Participant experienced at least 2 colds per year in the last 12 months

Exclusion Criteria:

1. Chronic respiratory tract or lung disease (e.g. chronic bronchitis, COPD, bronchial asthma, cystic fibrosis, active pulmonary tuberculosis, lung cancer)
2. History of heart, renal, liver, neuromuscular disease and/or immunosuppression
3. Known allergic bronchial asthma
4. Known or suspected congenital anomalies of heart, kidney, liver, or mental disabilities
5. Participant with concomitant medications that might impair the interpretation of trial results (e.g. herbal medications for common cold other than the investigational product, or pain relief medications other than Paracetamol or Ibuprofen)
6. Women of child-bearing potential with no adequate and effective contraception (MHRA, 2010):

   * Established use of oral, injected or implanted hormonal methods of contraception
   * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
   * Barrier methods of contraception: Condom and/or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
   * Sexual abstinence
   * Vasectomised partner
7. Female participant who is pregnant, lactating or planning pregnancy during the course of the clinical trial
8. Participant with cold symptoms at inclusion
9. Current intake of antimicrobial and/or antiviral medication for any reason
10. Participant with known or suspected history of alcohol or drug abuse
11. Heavy smoking (more than 10 cigarettes per day)
12. Psychiatric disorders which may influence the results of the trial, epilepsy, or suicide attempts
13. Planned surgical intervention during the trial
14. Known gastrointestinal disorders with uncertain absorption of orally administered medication (e.g. partial or total gastrectomy, enterectomy, inflammatory bowel disease, celiac disease, symptomatic lactose intolerance, dysbacteriosis) or associated with diarrhoea
15. Known or suspected hypersensitivity to the active substance or to any of the excipients of the investigational product
16. Known clinically relevant laboratory abnormalities
17. Participant with increased tendency to bleed, especially nasal or gingival bleeding
18. Previous (within the last 3 months prior to visit 1) or concomitant treatment with coagulation-inhibiting drugs such as warfarin
19. Participation in a further clinical trial at the same time or within the last 4 weeks prior to inclusion into the present study
20. Previous randomisation in the present clinical study
21. Irresponsible subjects or those unable to understand nature, meaning and consequences of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse Drug Reactions (ADRs) | during the 4 months treatment

SECONDARY OUTCOMES:
Occurrence of Adverse Events (AEs) during the 4 months treatment | Adverse events will be documented during the 4 months treatment period.
Protective effects | Protective effects will be evaluated during the 4 months treatment period.
  Time to onset of first common cold symptoms, time between last common cold episode prior to trial entry and first cold episode during the trial, total number of common cold episodes, total number of participants with at least one / more than one common cold episode
Effects during a cold episode | Treatment effects on common cold symptoms will be documented for 14 days after onset of first common cold symptom
  Mean cold episode duration (in days), cumulative episode days, number of co-medicated cold episodes, number of patients with respiratory complications due to common cold, development of the total cold symptom score and of single symptoms during a cold episode

CONTACTS AND LOCATIONS:
Overall Officials: Moutaz SM Jawad, M.B., B.Ch., FRCP, Principal Investigator — Common Cold Centre, Cardiff School of Biosciences, Cardiff University
Locations (1):
- Cardiff University, Common Cold Centre, Cardiff School of Biosciences, Cardiff, Wales, United Kingdom